CLINICAL TRIAL: NCT07040124
Title: Assessment of Efficacy of Prebent Titanium Mesh Versus Customized Poly-ether Ether Ketone Mesh for Three Dimensional Augmentation in Deficient Maxillary Ridge. a Randomized Controlled Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basma Alsheikh (Other)
Responsible Party: Sponsor-Investigator, Basma Alsheikh, assistant lecturer, British University In Egypt
Organization: British University In Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1125486
Record Dates: First submitted 2025-06-25; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Deficient Alveolar Bone
Keywords: augmentation,; peek; titanium mesh

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prebent titanium mesh (Active Comparator): participants receive alveolar ridge augmentation using pre-bent titanium mesh
  Interventions: Procedure: ti mesh
- 3d peek mesh (Active Comparator): participants receive maxillary ridge augmentation using 3d milled peek mesh
  Interventions: Procedure: 3d peek mesh

INTERVENTIONS:
Procedure: ti mesh — prebent titamesh on a 3-d virtually augmented model
  Arms: prebent titanium mesh
Procedure: 3d peek mesh — milled 3d peek mesh
  Arms: 3d peek mesh

SUMMARY:
In conclusion, the choice between titanium and PEEK meshes should consider patient-specific factors, clinical requirements, and surgeon expertise. The PEEK mesh, with its patient customized design enabled by CAD/CAM technology, offers significant advantages, including greater gained bone volume and reduced operative time. Its tailored fabrication ensures precise adaptation to the patient's anatomy, effectively maintaining the space required for optimal bone formation. The integration of such advanced technologies in regenerative procedures represents a significant step forward in achieving predictable outcomes and enhancing patient care. However, continued innovation and evaluation are crucial to refine these approaches and expand their applicability in oral rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patient of both sexes presenting with partially edentulous maxillary ridge with horizontal bone defect. 2. The horizontal ridge dimension measured 2mm below the alveolar crest should range from 2-5 mm. 3. No local pathosis that may interfere with bone healing. 4. Good oral hygiene. 5. Age between 20-65 years old.

Exclusion Criteria:

* Patient taking any medication that may interfere with normal bone physiology or impair bone healing. 2. All patients suffering from any systemic disease that may affect bone healing. 3. Heavy smokers (more than 10 cigarette per day) 4. Patients with parafunctional habits such as bruxism and clenching 5. Poor interest and cooperation from the patient. 6. Patients that have undergone any horizontal augmentation procedure at the site of interest

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
horizontal bone gain | 6 months
  cbct analysis for bone gain

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal Univresity, Suez, Egypt

IPD SHARING:
Plan to Share IPD: No